CLINICAL TRIAL: NCT04463537
Title: The Effect Of Auricle Position On Body Temperature Measurements Made With Tympanic Membrane Thermometer In Adults
Brief Title: The Effect of Auricle Position on Tympanic Thermometry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Nilay Orkun, Research Assistant (Phd), Ege University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-106
Record Dates: First submitted 2020-07-07; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Body Temperature Changes
Keywords: body temperature,; adult patients,; tympanic membrane thermometer,; auricle position,; nursing practice.
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Intervention Model Description: a quasi-experimental design with a pre-test and a post-test.
Masking Description: A total of 143 patients who fit the inclusion criteria of the study were included in the sample. The research carried out between 1 November - 31 December 2016 in the emergency department. Body temperature measurements were carried out on the patients in the study firstly by not changing the position of the auricle and then repeated after a minute, this time by changing the position of the auricle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experiment group (Experimental): Firstly, patients selected with convenience sampling. In the sampling method, the order of the patients' enrollment to the emergency room was used. Then, patient's age, sex and presence of otitis media were recorded in the Personal Information Form.
  After recording, measurements were carried out on the patients in the study firstly by not changing the position of the auricle. The duration was measured by stop watch and the results were recorded in the data form. The levels of patients' discomfort were evaluated by the "Visual Comparison Scale".
  The measurement was then repeated after a minute, this time by changing the position of the auricle. The duration was measured for this position and the results were recorded in the data form. The levels of patients' discomfort were evaluated by the "Visual Comparison Scale". The auricle on the same side was used during both measurements.
  Interventions: Procedure: Body Temperature Measurements

INTERVENTIONS:
Procedure: Body Temperature Measurements — measurements were carried out on the patients in the study firstly by not changing the position of the auricle. The duration was measured by stop watch and the results were recorded in the data form. The levels of patients' discomfort were evaluated by the "Visual Comparison Scale".
  The measurement was then repeated after a minute, this time by changing the position of the auricle. The duration was measured for this position and the results were recorded in the data form.

SUMMARY:
Objective: The aim of this study was to investigate the effect of auricle position on body temperature measurements made with tympanic membrane thermometer in adult patients.

Methods: The study was conducted with a quasi-experimental design with a pre-test and a post-test. A total of 143 patients who fit the inclusion criteria of the study were included in the sample. The research carried out between 1 November - 31 December 2016 in the emergency department. Body temperature measurements were carried out on the patients in the study firstly by not changing the position of the auricle and then repeated after a minute, this time by changing the position of the auricle.

Results: The difference between the measurement values found in two different positions was 0.31 0C, and the Bland Altman plot showed that the differences were distributed systematically around the value 0.31. The difference between the lengths of measurements performed on two separate positions was detected to be 1.08 second. During body temperature measurements performed through giving position to auricle, 59.2 % of the patients never felt discomfort.

Conclusions: It was found in the comparison of two positions that there was a significant difference between the tympanic membrane thermometer measurements made by positioning the auricle and those without positioning.

DETAILED DESCRIPTION:
Introduction One of the most common practices in clinical investigations is the measurement of a patient's body temperature (1-2,3). Body temperature measurement has a significant place in evaluation of clinical pictures and clinical monitoring (4). The issue at hand is that various temperature measurement modalities yield different results (2-4).

Although the accuracy of temperatures measured by infrared tympanic thermometers is a controversial issue among people interested in the subject, these thermometers have many advantages; they measure the temperature fast (1-2 s), and they are easy to use and non-invasiveness (3). Compared to the armpit or oral temperatures, the tympanic temperature reﬂects the core temperature more accurately which was demonstrated by comparing the temperature measurements made in the pulmonary artery and esophagus (5-6).

Methods Aim The aim of this study investigate the effects of auricle position on body temperature values in tympanic membrane thermometer measurements performed on adult patients. The hypothesis was "Position of the auricle during measurement of tympanic membrane temperature will affect the reading".

Design The study was conducted with a quasi-experimental design with a pre-test and a post-test.

The Study Participants This cross-sectional study surveyed 143 patients from one of emergency department in Turkey. The patients who were 18 years old or older, conscious, without communication issues, volunteers, not diagnosed with otitis media, who did not have a fever. Because otitis media and fever cause to potential sources of bias. A sample of the study with 143 patients who meeting these criteria and agreed to participate in the study was generated.

Data collection The data were collected by "a Personal Information Form, a Visual Comparison Scale, a tympanic membrane thermometer and a stop watch" by the researcher on 143 patients who selected convenience sampling at the Emergency Services of a university hospital in the period of 1 November - 31 December 2016.

Data Collection Tolls The "Personal Information Form" is a form that includes three questions based on socio-demographic characteristics (age, sex, presence of otitis media), this form was developed by the researchers. "Tympanic membrane thermometer" were used during body temperature measurements. The "Visual Comparison Scale" is used in evaluating the discomfort the patients feel based on auricle position change during the body temperature measurement, and it records the values for the duration of the body temperature measurement process and body temperature. This form was developed by the researchers. The score range of the "Visual Comparison Scale" is between 0 and 10.

According to this scale, while "0" means "I do not feel discomforted", "10" means "I feel terribly discomforted". "Stop watch" was used to record whether there is a difference between the measurement processes in terms of duration.

To measure the body temperature in all the patients, only the Covidien brand tympanic membrane thermometer was used. Before the study was started, the Covidien brand tympanic membrane thermometer was calibrated and a pilot study was conducted with 15 people to assure the accuracy of the thermometer.

Intervention Firstly, patients selected with convenience sampling. In the sampling method, the order of the patients' enrollment to the emergency room was used. Then, patient's age, sex and presence of otitis media were recorded in the Personal Information Form.

After recording, measurements were carried out on the patients in the study firstly by not changing the position of the auricle. The duration was measured by stop watch and the results were recorded in the data form. The levels of patients' discomfort were evaluated by the "Visual Comparison Scale".

The measurement was then repeated after a minute, this time by changing the position of the auricle. The duration was measured for this position and the results were recorded in the data form. The levels of patients' discomfort were evaluated by the "Visual Comparison Scale". The auricle on the same side was used during both measurements.

Sample Size Calculation In order to determine the sample size, a pre-administration was conducted on a total of 15 adult patients. The collected data were subjected to a power analysis. The effect size was determined as d=0.3645, according to the evaluation that was conducted by using these data. To obtain 99% power at a level of α=0.05, it was determined that there must be 110 patient in the groups. When considering that there may be a loss of data in the study process, it was decided that the study should be conducted on a total of 143 participants.

Ethical Considerations Approval (number: 2015-106) was received for the study from the Scientific Ethics Board of University, Faculty of Nursing. Written permission was taken from the Chief Physician of the Hospital of University, Faculty of Medicine for conducting the study in the emergency department of the hospital, while written consent was received from patients themselves after information was provided about the purpose of the study.

Analysis The statistical analysis of the data obtained in the study was achieved using the Statistical Package for the Social Sciences (SPSS) 22.0. For analysis of the data, frequencies, percentages, means and standard deviations were calculated, and the significance of the difference between paired values was tested in order to investigate the effects of auricle position on measurement values. Additionally, systematic distributions of the data were examined with a Bland Altman plot which is used in repeated measurements based on positions. The results were interpreted in a 95% confidence interval and a level of significance of p<0.05.

The mean value taken from the measurements with the tympanic membrane thermometer was 36.99±0.48 in measurements by positioning the auricle, and 36.68±0.47 in measurements without positioning. The difference between the measurements obtained in two different positions was found as 0.31 0C. Accordingly, it was found that the difference between the values in two different measurement positions was noteworthy (t=15.12; p< 0.05).

While one of the researchers measured the temperature with the tympanic membrane thermometer, the other researcher measured the amount of time elapsed with a stopwatch and recorded it. The mean duration of measurement was 5.51 seconds (min: 3.5 max: 7.3) in the measurements made by positioning the auricle, and 4.42 seconds (min: 2.9 max: 7.6) in the measurements without positioning. Considering the difference between the durations of measurements made in two different positions ( =1.08±0.07) it was found that the difference was significant between the measurements with positioning and those without positioning (t=15.16; p< 0.05).

Table II. Measurement results according to pinna position and durations of the measurements taken in the comparison of the two positions.

Conclusion This article contributes the main finding that nurses should be change the position of the pinna while measuring the temperature with tympanic membrane thermometers. Placing the sensor tip of the thermometer into the ear canal and pulling the auricle allows easy access to the tympanic membrane by straightening the external canal and it reflected the core temperature accurately.

Utilization of tympanic membrane thermometers in measurement of body temperature is highly important and technique should be applied properly to obtain correct values in emergency department. In the light of the results we obtained in this study, in order to achieve accurate and reliable measurement values the auricle should be positioned correctly, and the ear canal should be straightened. This way, the tympanic membrane that receives blood via the external cerebral artery is placed straight ahead the infrared rays. This method of body temperature measurement should be included in the in-service training or nurses, as it is one of the jobs of nurses to measure body temperature.

The information in user manuals in Turkish about tympanic membrane thermometers should be updated to include the steps in the process of body temperature measurement, and nurses should use this method effectively. The information in the literature relative to nursing practices on measurements made with tympanic membrane thermometers should be updated. It was found that the measurements made by positioning the auricle did not require an extra application time and this application would not be an additional workload for the nurses. It was determined that body temperature measurement by placing auricle in position did not cause discomfort in patients. Studies about the accuracy and reliability of measurements made with tympanic membrane thermometers should be repeated on different samples and the results should be shared.

References

1. Chaglla JSE, Celik N, Balachandran W. Measurement of Core Body Temperature Using Graphene-Inked Infrared Thermopile. Sensor 2018;18:3315-23. Doi: 10.3390/s18103315.
2. Arslan GG, Eşer İ, Khorshıd L. Analysis of the effect of lying on the ear on body temperature measurement using a tympanic thermometer. Journal of Pakistan Medical Association 2011; 61:1065. Retrieved from http://jpma.org.pk/PdfDownload/3100.pdf.
3. Erickson RS, Kirklin SK. Comparison of ear-based, bladder, oral, and axillary methods for core temperature measurement. Critical care medicine, 1993;21(10): 1528-1534.
4. Yeoh WK, Lee JKW, Lim HY, Gan CW, Liang W, Tan KK. Re-visiting the tympanic membrane vicinity as core body temperature measurement site. PLoS ONE 2017; 2 (4): 1-21. Doi: 10.1371/journal.pone.0174120.
5. Stavem, Saxholm, Smith-Erichsen, 1997
6. Yaron M, Lowenstain SR, Koziol McLain J. Measuring the accuracy of the infrared tympanic thermometer. Journal of Emergency Medicine 1995;13:617-621. Doi: 10.1016/0736-4679(95)00065-i

ELIGIBILITY:
Inclusion Criteria:

The patients who were 18 years old or older, conscious, without communication issues, volunteers, not diagnosed with otitis media, who did not have a fever.

Exclusion Criteria:

havin fever, Being under the age of 18, not volunteers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-01-05 (Actual)

PRIMARY OUTCOMES:
outcome1 | NOVEMBER 2016 JANUARY 2017
  It was found in the comparison of two positions that there was a significant difference between the tympanic membrane thermometer measurements made by positioning the auricle and those without positioning

IPD SHARING:
Plan to Share IPD: No
I have not IPD